CLINICAL TRIAL: NCT00862329
Title: Influence of Protein Source on Satiety and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Manager of the HNRC, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SURPROL
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Healthy subjects
MeSH Terms: interventions — Caseins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Casein (Experimental)
  Interventions: Dietary Supplement: Casein-enriched diet
- MSP (Experimental)
  Interventions: Dietary Supplement: Milk soluble protein-enriched diet
- Casein/MSP (Experimental)
  Interventions: Dietary Supplement: Casein and milk soluble proteins-enriched diet
- Soy protein (Experimental)
  Interventions: Dietary Supplement: Soy proteins-enriched diet

INTERVENTIONS:
Dietary Supplement: Casein-enriched diet — Subjects consume for 9 days a supplement of 30g/d of casein
  Arms: Casein
Dietary Supplement: Milk soluble protein-enriched diet — Subjects consume for 9 days a supplement of 30g/d of milk soluble protein
  Arms: MSP
Dietary Supplement: Casein and milk soluble proteins-enriched diet — Subjects consume for 9 days a supplement of 30g/d of a mix of casein and milk soluble protein
  Arms: Casein/MSP
Dietary Supplement: Soy proteins-enriched diet — Subjects consume for 9 days a supplement of 30g/d of soy protein
  Arms: Soy protein

SUMMARY:
Dietary protein is the more satiating nutrient, however it is not clear whether satiety may be influenced by the nature of the protein. This study was designed to assess potential differences between protein sources on satiety and their relationship with digestive and metabolic kinetics.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 30

Exclusion Criteria:

* allergy to milk proteins

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
satiety | 7 days

SECONDARY OUTCOMES:
hormonal profiles, digestive fluxes of nutrients, postprandial dietary N metabolism | 9 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur volontaires, Bobigny, France

REFERENCES:
- [Derived] Marsset-Baglieri A, Fromentin G, Airinei G, Pedersen C, Leonil J, Piedcoq J, Remond D, Benamouzig R, Tome D, Gaudichon C. Milk protein fractions moderately extend the duration of satiety compared with carbohydrates independently of their digestive kinetics in overweight subjects. Br J Nutr. 2014 Aug 28;112(4):557-64. doi: 10.1017/S0007114514001470. Epub 2014 Jun 26. PMID 24968280
- [Derived] Boutrou R, Gaudichon C, Dupont D, Jardin J, Airinei G, Marsset-Baglieri A, Benamouzig R, Tome D, Leonil J. Sequential release of milk protein-derived bioactive peptides in the jejunum in healthy humans. Am J Clin Nutr. 2013 Jun;97(6):1314-23. doi: 10.3945/ajcn.112.055202. Epub 2013 Apr 10. PMID 23576048